CLINICAL TRIAL: NCT06638008
Title: Ultrasound Guided Placental Growth Factor Vs Platelet Rich Plasma Injection in Peripheral Nerve Injury: an Interventional Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Taher Mohamed Amin, Main investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sara thesis
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Nerve Injury Upper Limb
Keywords: peripheral nerve injury; median and ulnar nerves; nerve conduction study; neuromuscular ultrasound; placental growth factor; perineural injection; platelet rich plasma
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group will receive placental growth factor injection (Experimental)
  Interventions: Drug: perineural injection
- group will receive platelet rich plasma injection (Experimental)
  Interventions: Drug: perineural injection
- group with only follow up (No Intervention)

INTERVENTIONS:
Drug: perineural injection — perineural intervention of placental growth factor in one group and PRP in other group
  Arms: group will receive placental growth factor injection; group will receive platelet rich plasma injection

SUMMARY:
The goal of this clinical trial is to learn if placental growth factor injection and platelet rich plasma injection works to treat peripheral nerve injury in adults. and the role of nerve conduction study and neuromuscular ultrasound

The main questions it aims to answer are:

Does placental growth factor improve outcome after peripheral nerve injury? Does platelet rich plasma improve outcome after peripheral nerve injury? Researchers will compare drug both drugs to each other and will follow up the results via NCS and NMUS

Participants will be classified into 3 random groups:

one group will receive perineural injection of placental growth factor, the other group will receive peri neural PRP injection, third group will only be followed up without intervention Follow up of each patients will be done at 3 and 6 months

DETAILED DESCRIPTION:
Traumatic nerve injuries, particularly involving the median and ulnar nerves, pose significant clinical challenges and can lead to considerable morbidity Neuropathic pain, which can arise from nerve lesions, may persist for months or even years after the apparent healing of the affected tissues , Moreover, weakness or paralysis of specific muscles can impair grip strength and fine motor skills, making daily tasks challenging, and the chronic disability affects patient's quality of life.

Neuromuscular US is a non-invasive technique to diagnose peripheral nerve injuries, basic findings in nerve trauma may include focal enlargements suggesting a neuroma in continuity, disorganization of the internal fascicular structure, as well as partial or complete nerve transection.

Growth factors play a pivotal role in the process of nerve regeneration by promoting cellular growth, survival, and differentiation.

Placenta extract contains a variety of growth factors, such as: Vascular Endothelial Growth Factor (VEGF), Transforming Growth Factor-beta (TGF-β), Fibroblast Growth factor (FGF) and insulin-like growth factor (IGF), It also includes cytokines and proteins that support healing and modulate inflammatory responses(6)placental extract use showed a significant improvement in pain and range of motion in knee osteoarthritis, Fibromyalgia and Rheumatoid arthritis (RA).

Another rich source of growth factors is platelet-rich plasma (PRP) it allows gradual and sustained release of neurotrophic signaling molecules such as nerve growth factor (NGF), Brain-Derived Neurotrophic Factor (BDNF), IGF-1, platelet-derived growth factor (PDGF), VEGF, and hepatocyte growth factor (HGF) and neurotropic factors (fibrin, fibronectin, and vitronectin) Studies on PRP and placental extract effect on nerve injuries are also still limited which needs further experimentation to understand its effect, and ability of regeneration of various neural components.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients older than 16 yrs old.
2. Patients with traumatic median or ulnar nerve injury who are complaining of symptoms or functional disability.
3. Patients with these injuries for more than 3 months

Exclusion Criteria:

* 1- Presence of other causes of nerve affection (entrapment, Diabetes, etc).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of placental growth factor injection guided by ultrasound and nerve conduction | one year
  pre and post injection follow up will be done my measuring the nerve conduction velocity and amplitude , and by determining the cross sectional area of the nerve by ultrasound
efficacy of platelet rich plasma injection guided by ultrasound and nerve conduction | one year
  pre and post injection parameters of nerve conduction as velocity and amplitude will be measured as will as parameters of ultrasound such as cross sectional area

SECONDARY OUTCOMES:
diagnosis and follow up of patients by nerve conduction study and neuromuscular US | one year
  patients will undergo baseline NCS and NMUS and then follow up the outcome of injection at 3 and 6 months the following parameters will be measured : nerve conduction velocity and amplitude as well as cross sectional area of the nerve

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ahmed Abda, professor, Principal Investigator — professor of Rheumatology, Rehabilitation and physical medicine; Mohammed Raouf Abd El-razik, Assistant professor, Study Director — Assistant professor of Rheumatology, Rehabilitation and physical medicine; Amira Mostafa El-sonbaty, lecturer, Study Director — lecturer of Rheumatology, Rehabilitation and physical medicine

IPD SHARING:
Plan to Share IPD: Undecided